CLINICAL TRIAL: NCT01183832
Title: Radiotherapy - Anastrazole Concomitant : Evaluation of the Side Effects
Acronym: ORACLES
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: ORACLES
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; radiotherapy; hormonotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concomitant: In this group, anastrazole is concomitant to the radiotherapy
- Sequential: In this group, anastrazole is sequential to the radiotherapy (start after the end of radiotherapy)

SUMMARY:
This study is a description of the radiation effects on the healthy tissues in patients receiving Anastrozole, sequential or in association with radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal woman without superior age limit
* No metastatic breast cancer, stade I-II, estrogen receptor positive or progesterone receptor positive, treated by conservative surgery or total mastectomy and requiring additive treatment by radiotherapy and hormonotherapy
* The patients including in another clinical trial can be include in this observatory

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are post-menopausal women treated for a breast concer
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2005-08; Primary Completion 2015-01-13 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
radiation side effects | 5 years after the end of radiotherapy
  Describe, in real situation, the ionisant radiation effects on the healthy tissues in patients receiving anastrazole in association or sequential with radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Yazid BELKACEMI, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (29):
- France (28):
  - Centre Henri Becquerel, Amiens
  - Clinique La Casamance, Aubagne
  - Hôpital Duchêne, Boulogne-sur-Mer
  - Centre François Baclesse, Caen
  - Charleville
  - Henri Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Clinique Clairval, Marseille
  - Institut Paoli Calmettes, Marseille
  - La Timone, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Hospitalier St Grégoire, Nantes
  - Nouvelles cliniques nantaises, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Antoine LACCASSAGNE, Nice
  - Clinique de la Roseraie, Paris
  - Hôpital Européen Georges Pompidou HEGP, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier LYON Sud, Pierre-Bénite
  - Polyclinique de Courlancy, Reims
  - Centre: Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Centre de radiothérapie Saint-Louis, Toulon
  - Centre Claudius REGAUD, Toulouse
  - Institut Gustave Roussy, Villejuif
- Centre CHPG, Monaco, Monaco